CLINICAL TRIAL: NCT03523286
Title: Real-time Automated Program for IDentification of VT Origin - Pilot Study
Brief Title: Real-time Automated Program for IDentification of VT Origin
Acronym: RAPIDVTPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amir AbdelWahab (Other)
Collaborators: Maritime Heart Centre (Other)
Responsible Party: Sponsor-Investigator, Amir AbdelWahab, Attending Cardiac Electrophysiologist, Associate Professor of Medicine, Division of Cardiology, Department of Medicine, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6201
Record Dates: First submitted 2018-04-09; First posted 2018-05-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Ventricular Tachycardia; Ischemic Heart Disease
Keywords: Catheter ablation; ECG imaging
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAPID-VT Software guided ablation (Experimental): The induced VT(s) 12-lead ECG will be acquired by the RAPID-VT software which will provide real time localization of the VT(s) exits from the scar margin. These exits will be targeted by ablation
  Interventions: Other: RAPID-VT Software guided ablation

INTERVENTIONS:
Other: RAPID-VT Software guided ablation — Catheter ablation will target VT exit sites at scar margin as determined by the RAPID-VT software

SUMMARY:
RAPID-VT Pilot is a single centre prospective cohort pilot study to assess the feasibility, safety and efficacy of catheter ablation of ventricular tachycardia (VT) guided by a novel real-time software to localize the origin of VT during the ablation procedure.

DETAILED DESCRIPTION:
Consecutive patients with ischemic heart disease and clinical indication of VT ablation will undergo baseline clinical evaluation, echocardiography and cardiac CT imaging using a contrast-enhanced cardiac-gated method with a 64-section scanner. Trans-axial CT images comprising the whole heart volume will be exported in DICOM format. CT image processing will be performed and will be used to delineate the LV endocardial and/or epicardial geometries. These data will be imported into the RAPID-VT software and the 3D-electranatomical mapping system for image integration.

During the VT ablation procedure, VT(s) induction will be performed. The VT(s) 12-lead ECG will be acquired by the RAPID-VT software and will be localized to the scar margin using the RAPID-VT software. Catheter ablation will be attempted at software-determined sites.

Post procedure, patient will be followed up for a minimum of 6 months. That will include Remote ICD follow-up and telephone study visits. Follow-up at 6 months will include a clinic visit for assessment of heart failure status, ECG, ICD interrogation and changes in antiarrhythmic drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion if they fulfilled VANISH inclusion criteria by having both of:

  1. Prior myocardial infarction (pathological Q waves or imaging evidence of regional myocardial akinesis/thinning in the absence of a non-ischemic cause)38 and
  2. One of the following VT events within the last 6 months while on Amiodarone or another class III or class I antiarrhythmic drug:

A: Sustained monomorphic VT documented on 12-lead ECG or rhythm strip requiring termination by pharmacologic means or DC cardioversion, B: ≥3 episodes of symptomatic VT treated with anti-tachycardia pacing (ATP), C: ≥1 appropriate ICD shocks, D: ≥3 VT episodes within 24 hours, separated by ≥ 5 minutes, E: sustained VT below detection rate of an ICD

Exclusion Criteria:

* Patients will be excluded from the trial if they:

  1. Are unable or unwilling to provide informed consent.
  2. Have active ischemia or another reversible cause of VT (e.g. drug-induced arrhythmia), or had recent acute coronary syndrome requiring revascularization.
  3. Are antiarrhythmic drug-naïve.
  4. Are known to have protruding left ventricular thrombus or mechanical aortic and mitral valves.
  5. Have had a prior catheter ablation procedure for VT.
  6. Are in renal failure (Creatinine clearance <15 mL/min)
  7. Have NYHA Functional class IV heart failure or CCS Functional class IV angina.
  8. Have had recent ST elevation myocardial infarction (< 1 month).
  9. Are pregnant or have a systemic illness likely to limit survival to <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Non-inducibility of VT | At end of ablation procedure
  Lack of any inducible VT at the end of the ablation procedure

SECONDARY OUTCOMES:
Procedure efficacy measure: VT(s) ablated | At end of procedure
  Number of VTs identified and targeted with ablation
Procedure efficacy measure: Procedure duration | At end of procedure
  Duration of procedure in minutes
Procedure efficacy measure: VT recurrence | During follow up period of 6 months
  Time to recurrence of VT in months
Procedure safety measure: Acute complications | At end of procedure and at 30 days of follow up
  Incidence of any procedure-related complications
Procedure safety measure: Clinical heart failure worsening | At end of procedure, at 30 days and 6 months of follow up
  Worsening of heart failure symptoms as defined as decline in NYHA Functional class or 6-MWT
Procedure safety measure: Mortality and hospitalization for cardiac causes | At 30 days and 6 months of follow up
  Death and/or cardiac hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Amir AbdelWahab, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- QE II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No